CLINICAL TRIAL: NCT03249805
Title: Efficacy of a New Design of Foot Abduction Brace (FAB) Compared to Standard FAB During Ponseti Treatment of Idiopathic Clubfoot by Measuring Rate of Recurrence and Compliance Using Novel Touch Sensors
Brief Title: MiracleFeet Foot Abduction Brace Sensor Trial
Acronym: mFAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MiracleFeet (Other)
Collaborators: Bai Jerbai Wadia Hospital for Children, Mumbai, India (Unknown); Metwiz Materials (Unknown); CURE (Unknown); Biomedical Engineering and Technology (Incubation) Center, Bombay (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2017-07-27; First posted 2017-08-15 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Clubfoot; Telemedicine; Patient Compliance
Keywords: LMIC; Medical device efficacy
MeSH Terms: conditions — Clubfoot; Patient Compliance

STUDY DESIGN:
Intervention Model Description: This will be a hospital-based study with single blinding of the investigator. Subjects will be randomized in order to prevent systematic differences between the groups to prevent bias. Our groups will be parallel, there will be no crossover. The two parallel groups will use two different versions of FABs; the Steenbeek Foot Abduction Brace (SFAB) and the MiracleFeet Foot Abduction Brace (mFAB). Both types of FAB will be equipped with discretely hidden sensors; subjects and their families will not be aware of the actual function of the sensor to avoid increased compliance due to the sensor. Due to practical constraints (the brace being visibly identifiable), the study will not be blind. This study will use number of recurrences in the two groups as the primary outcome of interest. Recurrence will be checked for at each scheduled follow-up visit (see schedule below) and recorded in event of occurrence. A process of rolling recruitment will be used until our groups are complete.
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Steenbeek Foot Abduction Brace (SFAB) (Experimental): The study will follow the subject for 6 months after their enrollment, beginning at first FAB use. The Steenbeek Foot Abduction Brace (SFAB) is a fixed metal bar attached to two leather shoes with laces. The shoes have laces and a strap. The FABs provide 10 degrees of dorsiflexion and 45 or 65 degrees of abduction, and will be equipped with sensors to measure at-home FAB compliance. After the last cast is removed, a brace will be worn for 23 hours/day for the first 3 months and the time will be gradually decreased thereafter to a 'nights and naps' protocol for a total of 12 hours/day. At follow-up appointments the brace will be checked for fit and Pirani score recorded.
  Interventions: Device: Steenbeek Foot Abduction Brace (SFAB)
- MiracleFeet Foot Abduction Brace (mFAB) (Experimental): The study will follow the subject for 6 months after their enrollment, beginning at first FAB use. The MiracleFeet Foot Abduction Brace (mFAB) is an injected plastic molded bar with fabric shoes that clip off and on. The shoes have laces and a strap. Both FABs provide 10 degrees of dorsiflexion and 45 or 65 degrees of abduction, and will be equipped with sensors to measure at-home FAB compliance. After the last cast is removed, a brace will be worn for 23 hours/day for the first 3 months and the time will be gradually decreased thereafter to a 'nights and naps' protocol for a total of 12 hours/day. At follow-up appointments the brace will be checked for fit and Pirani score recorded.
  Interventions: Device: MiracleFeet Foot Abduction Brace (mFAB)

INTERVENTIONS:
Device: Steenbeek Foot Abduction Brace (SFAB) — The FAB will be equipped with discretely hidden sensors; subjects and their families will not be aware of the actual function of the sensor in order to avoid increased compliance due to the sensor. Sensors work on the principle of force-sensing resistor material whose resistance changes when a force or pressure is applied. Force-sensing resistors consist of a conductive polymer, which changes resistance in a predictable manner following application of force to its surface. On the top of braces sole we have fixed force resistive sensor (FSR), which changes resistance whenever force is applied. Threshold of detection is 30-40 gram. The changes of resistance is detected by using micro-controller.
  Other Names: Denis Browne splint
  Arms: Steenbeek Foot Abduction Brace (SFAB)
Device: MiracleFeet Foot Abduction Brace (mFAB) — Sensors in the mFAB will measure whether the shoe is on, the foot is in contact with the sole of the shoe and the shoes are clipped into the bar. Sensors work on the principle of force-sensing resistor material whose resistance changes when a force or pressure is applied. Force-sensing resistors consist of a conductive polymer, which changes resistance in a predictable manner following application of force to its surface. On the top of braces sole we have fixed force resistive sensor (FSR), which changes resistance whenever force is applied. Threshold of detection is 30-40 gram. The changes of resistance is detected by using micro-controller.
  Other Names: Denis Browne splint
  Arms: MiracleFeet Foot Abduction Brace (mFAB)

SUMMARY:
The aim of this study is to determine the effect of a new design of FAB type on compliance and treatment outcomes of idiopathic clubfeet treated by the Ponseti method. Very little literature exists on the effect of brace type or the difference between reported and actual at-home compliance, which is integral to the success of treatment with the Ponseti method. Eighty children less than 1 year of age will be enrolled in the study into two arms, using block randomization. These two groups will use two different designs of foot abduction brace (FAB). Outcomes will be measured by number of recurrences per group (using recasting and/or surgical procedures and Pirani score as indicators), time of recurrences (in months), compliance with brace wear using sensors and comparing the data with brace wear reported by parents, and parent satisfaction with FAB (measured on a modified Orthotics and Prosthetics User Sur vey). Enrollment will be on a rolling basis; subjects will be enrolled at their last cast application and followed for approximately 6 months. Recurrences, time of recurrence, parent satisfaction, and reported vs. actual compliance will be analyzed.

DETAILED DESCRIPTION:
Clubfoot is the most common birth defect affecting 1 in every 750 live births, that is about 200,000 babies each year globally (80% mainly in developing countries). An estimated average 1 million children are currently living with untreated clubfoot. In India every 10 minutes a child is born with clubfoot i.e. over 50,000 children are born with this deformity every year (1 per 500 birth). The Ponseti Method is now recognized as the accepted standard for the medical treatment of clubfoot. The Ponseti Method is ideally suited for the developing world in that it is inexpensive, non-surgical and the casting component can be completed by trained medical and paramedical personnel. Clubfoot causes the feet of the affected individual to point downward and inward. Left untreated, clubfoot causes a permanent physical disability, preventing the individual from walking normally and limiting his or her mobility. Decreased ambulation can lead to the inability to perform daily tasks, such as going to school, leading to increased dependency and a negative economic impact on the family. Furthermore, deformity caused by neglected clubfoot can lead to limited social integration and stigma for both the individual and the family.

The gold standard of clubfoot treatment is the Ponseti method, which consists of 6-8 weeks of serial castings followed by a percutaneous Tendo Achilles tenotomy in the majority of cases. The casting is followed by the use of a foot abduction brace (FAB) for approximately 4 years. The goal of the treatment is to correct the deformity so that the patient has a functional, painless, plantigrade foot with full mobility without the need for orthotics. The 6-8 weeks of serial casting corrects the clubfoot deformity while the use of the FAB after casting prevents the deformity from reoccurring and is required for successful treatment. Noncompliance of FAB use increases the risk of relapse 17-fold.

Currently, the Steenbeek Foot Abduction Brace (SFAB), a version of the Denis Browne splint, is the only low-cost FAB available. The SFAB is made by hand by artisans, limiting its large-scale production. Furthermore, it can be challenging to put on a child due to the shoes being attached to the bar and lacking a strap in addition to laces, potentially leading to noncompliance.

The more recently developed MiracleFeet Foot Abduction Brace (mFAB) is made of injection molded plastic, making it easy to mass produce, and includes removable shoes with a strap to hold the heel in place, claiming to be more comfortable and easier to use, leading to improved compliance.

The MiracleFeet Foot Abduction Brace (mFAB) is a Denis Browne Splint used for the treatment of clubfoot. Use of the Denis Browne Split is standard in clubfoot treatment and the mFAB complies with the standards for foot abduction braces for clubfoot:

* Adjustable to 65 and 45 degrees to accommodate unilateral and bilateral clubfoot
* 10 degrees dorsiflexion

The mFAB was designed with the following additional features, based on requests from parents and providers:

* Large window to view the heel, ensuring it lays flat in the shoe
* Dorsal strap to secure the heel, allowing the shoe to be tied with two hands
* Removable shoes so that the shoes may be applied and then clipped into the bar
* A flat bottom
* The bar is made of strong injection-modeled plastic, in order to be reused
* The shoes are meant to be worn only by 1 child and then discarded

The mFAB shoes are made of canvas and polyester and the bar and shoe plates are made of ortholite and T90 and are manufactured using the injected-molded plastic process in Batavia, Illinois, USA.

The mFAB has been tested in Nicaragua, Brazil, South Africa and the Philippines and is currently in use in 10 countries. Both braces meet the specifications as detailed by the Ponseti method and the same bracing protocol is used for both.

This study will compare treatment outcomes and compliance using the two brace designs, SFAB and mFAB. We will compare the number and time of recurrences, as well as the reported compliance and actual compliance, which will be measured by novel sensors. Few studies exist that compare brace types or actual versus reported compliance and FABs with sensors are a novel technology. Of the literature that exists, FAB use was show to decline significantly during the first 3 months and actual wear is less than reported wear.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral cases of idiopathic clubfoot in children who have not yet started walking at first presentation, receiving a brace for the first time after successful correction with the Ponseti method of treatment, at the Bai Jerbai Wadia Hospital for Children over a period of 6 months.

Exclusion Criteria:

* All children who are already walking at presentation; All children with previous treatment; All children who have used FAB previously; All children treated with surgery other than tenotomy; All children with syndromic or neuropathic cases of clubfoot; All children with atypical clubfoot.

Ages: 3 Months to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2017-06-07 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Pirani Score | One year
  The Pirani score is a standardized tool measuring that severity of clubfoot deformity. It will be assessed at all visits - baseline, during treatment and follow-up - to evaluate gradual recurrence of clubfoot deformity.

SECONDARY OUTCOMES:
Orthotics Prosthetics User Survey (OPUS) Results | One year
  Parent satisfaction with the FABs will be determined by administering an OPUS to them at each follow-up visit.

OTHER OUTCOMES:
Minutes of brace usage per day | One year
  To measure at-home brace use compliance, the sensor data will be collected and compared to parent-reported brace usage. This will be tabulated in number of minutes the brace is used per day, collected at each follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Alaric Aroojis, MD, Principal Investigator — Bai Jerbai Wadia Hospital for Children
Locations (1):
- Bai Jerbai Wadia Hospital for Children, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ponseti IV. Treatment of congenital club foot. J Bone Joint Surg Am. 1992 Mar;74(3):448-54. No abstract available. PMID 1548277
- [Background] Morcuende JA, Dolan LA, Dietz FR, Ponseti IV. Radical reduction in the rate of extensive corrective surgery for clubfoot using the Ponseti method. Pediatrics. 2004 Feb;113(2):376-80. doi: 10.1542/peds.113.2.376. PMID 14754952
- [Background] Morgenstein A, Davis R, Talwalkar V, Iwinski H Jr, Walker J, Milbrandt TA. A randomized clinical trial comparing reported and measured wear rates in clubfoot bracing using a novel pressure sensor. J Pediatr Orthop. 2015 Mar;35(2):185-91. doi: 10.1097/BPO.0000000000000205. PMID 24787312
- [Background] Zionts LE, Frost N, Kim R, Ebramzadeh E, Sangiorgio SN. Treatment of idiopathic clubfoot: experience with the Mitchell-Ponseti brace. J Pediatr Orthop. 2012 Oct-Nov;32(7):706-13. doi: 10.1097/BPO.0b013e3182694f4d. PMID 22955535
- [Background] Boehm S, Sinclair M. Foot abduction brace in the Ponseti method for idiopathic clubfoot deformity: torsional deformities and compliance. J Pediatr Orthop. 2007 Sep;27(6):712-6. doi: 10.1097/BPO.0b013e3181425508. PMID 17717477
- [Background] Chen RC, Gordon JE, Luhmann SJ, Schoenecker PL, Dobbs MB. A new dynamic foot abduction orthosis for clubfoot treatment. J Pediatr Orthop. 2007 Jul-Aug;27(5):522-8. doi: 10.1097/bpo.0b013e318070cc19. PMID 17585260
- [Background] Garg S, Porter K. Improved bracing compliance in children with clubfeet using a dynamic orthosis. J Child Orthop. 2009 Aug;3(4):271-6. doi: 10.1007/s11832-009-0182-9. Epub 2009 Jun 3. PMID 19495824
- [Background] Hemo Y, Segev E, Yavor A, Ovadia D, Wientroub S, Hayek S. The influence of brace type on the success rate of the Ponseti treatment protocol for idiopathic clubfoot. J Child Orthop. 2011 Apr;5(2):115-9. doi: 10.1007/s11832-010-0321-3. Epub 2010 Dec 24. PMID 22468155
- [Background] Janicki JA, Wright JG, Weir S, Narayanan UG. A comparison of ankle foot orthoses with foot abduction orthoses to prevent recurrence following correction of idiopathic clubfoot by the Ponseti method. J Bone Joint Surg Br. 2011 May;93(5):700-4. doi: 10.1302/0301-620X.93B5.24883. PMID 21511939
- [Background] Kessler JI. A new flexible brace used in the Ponseti treatment of talipes equinovarus. J Pediatr Orthop B. 2008 Sep;17(5):247-50. doi: 10.1097/BPB.0b013e32830cc3e5. PMID 19471177
- [Background] Sangiorgio SN, Ho NC, Morgan RD, Ebramzadeh E, Zionts LE. The Objective Measurement of Brace-Use Adherence in the Treatment of Idiopathic Clubfoot. J Bone Joint Surg Am. 2016 Oct 5;98(19):1598-1605. doi: 10.2106/JBJS.16.00170. PMID 27707845
- [Background] Thatipelli S, Arun A, Chung P, Etemadi M, Heller J, Kwiat D et al. Review of Existing Brace Adherence Monitoring Methods to Assess Adherence. Journal of Prosthetics and Orthotics. 2016;28(4):126-135.
- [Background] Manousaki E, Czuba T, Hagglund G, Mattsson L, Andriesse H. Evaluation of gait, relapse and compliance in clubfoot treatment with custom-made orthoses. Gait Posture. 2016 Oct;50:8-13. doi: 10.1016/j.gaitpost.2016.08.005. Epub 2016 Aug 7. PMID 27544063
- [Background] Chong DY, Finberg NS, Conklin MJ, Doyle JS, Khoury JG, Gilbert SR. Prospective evaluation of the use of Mitchell shoes and dynamic abduction brace for idiopathic clubfeet. J Pediatr Orthop B. 2014 Nov;23(6):501-4. doi: 10.1097/BPB.0000000000000090. PMID 25144885
- [Background] Thacker MM, Scher DM, Sala DA, van Bosse HJ, Feldman DS, Lehman WB. Use of the foot abduction orthosis following Ponseti casts: is it essential? J Pediatr Orthop. 2005 Mar-Apr;25(2):225-8. doi: 10.1097/01.bpo.0000150814.56790.f9. PMID 15718907
- [Background] Ramirez N, Flynn JM, Fernandez S, Seda W, Macchiavelli RE. Orthosis noncompliance after the Ponseti method for the treatment of idiopathic clubfeet: a relevant problem that needs reevaluation. J Pediatr Orthop. 2011 Sep;31(6):710-5. doi: 10.1097/BPO.0b013e318221eaa1. PMID 21841450
- [Background] Bouchoucha S, Smida M, Saied W, Safi H, Ammar C, Nessib MN, Ghachem MB. Early results of the Ponseti method using the Steenbek foot abduction brace: a prospective study of 95 feet. J Pediatr Orthop B. 2008 May;17(3):134-8. doi: 10.1097/BPB.0b013e3282fa5f0d. PMID 18391812
- [Background] Desai L, Oprescu F, DiMeo A, Morcuende JA. Bracing in the treatment of children with clubfoot: past, present, and future. Iowa Orthop J. 2010;30:15-23. PMID 21045966